CLINICAL TRIAL: NCT03653871
Title: The Effect of a Performing Arts Intervention on People With Dementia and Their Caregivers
Brief Title: Caregiver Study Dr. Phillips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Dr. Phillips Center for the Performing Arts (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1236971
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer Disease; Dementia; Caregiver; Performing Arts
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Performing arts instruction delivered 1 hour/week for 8 weeks.
  Interventions: Behavioral: Performing Arts Instruction
- Wait List Control (No Intervention): Control group. Performing arts instruction delivered upon completion of control period.

INTERVENTIONS:
Behavioral: Performing Arts Instruction — Professionally delivered performing arts curriculum
  Arms: Intervention

SUMMARY:
This study will examine whether a performing arts class will improve the well-being of primary unpaid caregivers of people with dementia

DETAILED DESCRIPTION:
This study used sample size analysis to determine the adequately sized intervention group and control group, well-defined statistical methodology, and a well-documented intervention that can be easily replicated. The intervention has been developed by Dr. Phillips Center for the Performing Arts leadership with assistance from AMS Planning & Research.

ELIGIBILITY:
Inclusion Criteria:

* Primary, unpaid caregiver of person with dementia OR
* Person with Dementia.
* Live independently in the community.
* Care recipient has a Functional Assessment Staging Test (FAST) Score of 4-6b.
* Caregiver does not display symptoms of emotional, cognitive, or mental impairment.
* Caregiver must be able to produce adequate saliva sample.
* Caregiver/care recipient can travel to program.
* Caregiver/care recipient agree to participate in all aspects of study intervention and assessments.
* Caregiver is 18 years of age or older.
* Care recipient is 65 years of age or older
* Access to home phone or mobile phone

Exclusion Criteria:

* Unable to understand either spoken and/or written English.
* Caregiver is a paid employee of care recipient's legally appointed representative

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change caregiver burden as measured by Zarit Burden Interview | Baseline to 22 weeks
  Zarit Burden Interview is a caregiver self-report measure. The Interview uses a 5 point Likert Scale (Never - 0, Rarely - 1, Sometimes - 2, Quite Frequently - 3, Nearly Always - 4). Score can range from 0- to 88. 0-21 - little or no burden, 21-40 mild to moderate burden, 41-60 moderate to severe burden, 61-88 severe burden. A lower score represents a better outcome.
Change caregiver resiliency as measured by Brief Resiliency Scale | Baseline to 22 weeks
  Brief Resilience Scale is a self report of items using a 5 point Likert Scale. Three of the items, the scale is as follows: (Strongly Disagree-1, Strongly Agree -5) For the remaining 3 items, the scale is reversed (Strongly Agree - 5, Strongly Agree 1) Score can range from 6-30 and is divided by 6. A higher score represents a better outcome.

SECONDARY OUTCOMES:
Determine if intervention helps recovery from agitation and disruptive behavior for caregivers as measured by salivary cortisol levels | Baseline to week 10
  Salivary cortisol level
Determine if intervention improves caregiver's perception of care recipient's quality of life as measured by Quality of Life - Alzheimer's Disease | Baseline to 22 weeks
  Quality of Life - Alzheimer's Disease is a self-report of items using a 4 point Likert Scale (Poor - 1, Fair - 2, Good - 3, Excellent - 4) The score ranges from 13-52. A higher score represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kim McManus, PhD, Principal Investigator — AdventHealth
Locations (1):
- Dr. Phillips Center for the Performing Arts, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. (2017). 10 facts on dementia. Retrieved March, 2017, from http://www.who.int/features/factfiles/dementia/en/
- [Background] Wimo A, Guerchet M, Ali GC, Wu YT, Prina AM, Winblad B, Jonsson L, Liu Z, Prince M. The worldwide costs of dementia 2015 and comparisons with 2010. Alzheimers Dement. 2017 Jan;13(1):1-7. doi: 10.1016/j.jalz.2016.07.150. Epub 2016 Aug 29. PMID 27583652
- [Background] Schulz R, Sherwood PR. Physical and mental health effects of family caregiving. Am J Nurs. 2008 Sep;108(9 Suppl):23-7; quiz 27. doi: 10.1097/01.NAJ.0000336406.45248.4c. PMID 18797217
- [Background] Cohen GD, Perlstein S, Chapline J, Kelly J, Firth KM, Simmens S. The impact of professionally conducted cultural programs on the physical health, mental health, and social functioning of older adults. Gerontologist. 2006 Dec;46(6):726-34. doi: 10.1093/geront/46.6.726. PMID 17169928
- [Background] Houston TK, Allison JJ, Sussman M, Horn W, Holt CL, Trobaugh J, Salas M, Pisu M, Cuffee YL, Larkin D, Person SD, Barton B, Kiefe CI, Hullett S. Culturally appropriate storytelling to improve blood pressure: a randomized trial. Ann Intern Med. 2011 Jan 18;154(2):77-84. doi: 10.7326/0003-4819-154-2-201101180-00004. PMID 21242364